CLINICAL TRIAL: NCT03190070
Title: Measurement of Renal Functional Reserve With Urinary Clearance of Cold Iothalamate Before and After an Oral Protein Load
Brief Title: Measurement of Renal Functional Reserve
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Sushrut S Waikar, Constantine L. Hampers, MD Distinguished Chair in Renal Medicine, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2016P002287
Record Dates: First submitted 2017-06-14; First posted 2017-06-16 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Kidney Diseases
Keywords: Renal reserve, physiological study, diagnostic testing
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Intervention Model Description: Physiological study to measure the change in glomerular filtration rate after an oral protein load
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): All study participants are in the same group and will have their kidney function measured twice, before and after ingestion of protein, 1 g/(kg body weight). The protein will be given in the form of the protein drink Liquacel (Global Health Products, Rochester, NY).
  Interventions: Dietary Supplement: Ingestion of protein

INTERVENTIONS:
Dietary Supplement: Ingestion of protein — Oral protein load as a physiological stimulus to temporarily increase glomerular filtration rate
  Other Names: Liquacel (Global Health Products, Rochester, NY)

SUMMARY:
Single arm physiological study to measure renal functional reserve as a biomarker of kidney function and health

DETAILED DESCRIPTION:
The investigators will measure glomerular filtration rate using urinary clearance of cold iothalamate before and after an oral protein load in patients with chronic kidney disease and healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18
2. Estimated GFR >30 mL/min/1.73m2

Exclusion Criteria:

1. Allergy to iothalamate, shellfish or iodine
2. Use of metformin or amiodarone
3. Inability to maintain a stable regimen of medications which affect GFR for > one week prior to participation (e.g. non-steroidal anti-inflammatory drugs, angiotensin converting enzyme inhibitors, angiotensin receptor blockers)
4. Use of medications which directly affect elimination of creatinine (e.g. cimetidine and trimethoprim)
5. Acute exacerbation of asthma or chronic obstructive pulmonary disease within 3 months requiring hospitalization or oral steroid therapy
6. Inadequate intravenous access
7. Severe anemia (Hct <21%)
8. Acute kidney injury (rise in creatinine to ≥1.5 times the previous baseline or by ≥ 0.3 mg/dL on most recent labs prior to enrollment)
9. History of contrast-induced nephropathy
10. Hyperthyroidism
11. Pheochromocytoma
12. Sickle cell disease
13. Urinary retention or incontinence
14. Status post organ transplant
15. Pregnancy or active breast feeding
16. Cognitive impairment with inability to give consent
17. Institutionalized status

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2017-07-12 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Change in glomerular filtration rate after ingestion of protein | Single full-day clinic visit: Repeated glomerular filtration rate measurements are to be performed over the course of the day at a single study visit for each participant.
  Short term-changes in the glomerular filtration rate will be measured before and after ingestion of oral protein

CONTACTS AND LOCATIONS:
Overall Officials: Sushrut Waikar, MD MPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Palsson R, Waikar SS. Renal Functional Reserve Revisited. Adv Chronic Kidney Dis. 2018 May;25(3):e1-e8. doi: 10.1053/j.ackd.2018.03.001. PMID 29793670